CLINICAL TRIAL: NCT01882855
Title: Effect of Music on Attention and Prospective Memory in Hepatic Encephalopathy
Status: Withdrawn | Type: Observational
Why Stopped: Dr. Sigal no longer with NYUMC
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: S12-03729
Record Dates: First submitted 2013-05-01; First posted 2013-06-20 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Cirrhosis; Hepatic Encephalopathy
MeSH Terms: conditions — Fibrosis; Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Hepatic encephalopathy (HE) is a potentially reversible, metabolically caused complication of acute or chronic liver diseases such as cirrhosis. Due to the diseased liver's inability to remove toxins such as ammonia, which is produced in the gastrointestinal tract, the ammonia accumulates in the brain and causes forgetfulness, confusion, disorientation, concentration and memory problems, changes in mood, decreased alertness and responsiveness, changes in sleep habits, muscle tremors and stiffness, speech impairments, uncontrollable movements, agitation.

This study will examine music as a possible external factor that could contribute to impairment in attention and progressive memory in cirrhotic patients while driving. Sustaining attention is important for learning and remembering new information, for e.g. keeping the car within lane and paying attention to cyclists and pedestrians. Prospective memory is the ability to remember to perform previously intended tasks at the appropriate time or occasion, for instance remembering the correct exit while driving on the highway. Impairment in any of these areas may result in serious consequences for patient with cirrhosis. There is evidence that some subsets of cirrhotic patients have a diminished ability to drive and significantly more motor vehicle crashes and traffic violations. In these patients, listening to music while driving may further jeopardize their driving ability, which in turn may lead to reduced quality of life and increased medical costs (from motor vehicle accidents).

This is a cross-sectional study designed to determine if there is any effect of listening to music on attention and prospective memory in patients with cirrhosis. For these purposes, subjects will be asked to come for one study visit, which will last approximately 2 hours. During this visit, subjects will undergo a series of screening procedures (consent, assignment of subject identification number, demographics, medical history, physical examination, vitals, height, weight, and eligibility assessment). If they are found eligible, subjects will undergo several neuropsychological assessments to measure any effect of music on attention and prospective memory. These assessments include including Number Connection Test (NCT), Digit Symbol Test (DST), Cambridge Prospective Memory Test (CAMPROMPT) and Inhibitory Control Test (ICT).

DETAILED DESCRIPTION:
Cirrhosis occurs when scar tissue replaces healthy liver tissue, partially blocking blood flow and preventing the liver's ability to control infections, removes bacteria and toxins from the blood, and to produce proteins to regulate blood clotting and bile to absorb fats and fat-soluble vitamins. With an estimated prevalence between five and ten percent, cirrhosis is the twelfth leading cause of death by disease, leading to 27,000 deaths per year. Heavy alcohol consumption and hepatotropic viruses (hepatitis B and C) are the major contributors to this disease's prevalence (NDDIC, 2003).

Hepatic encephalopathy (HE) is a potentially reversible, metabolically caused complication of acute or chronic liver diseases such as cirrhosis, which is characterized by neuropsychiatric abnormalities. Nearly 70% of cirrhotic patients experience mild levels of HE and approximately 30% of end-stage patients experience significant HE symptoms, many approaching coma (Mullen et al., 1999). Although the pathophysiology of HE is not yet clearly understood, the accumulation of ammonia in the brain due to the liver's inability to remove toxins (including ammonia) is thought to play a key role in the pathogenesis of HE. Other factors, which are not mutually exclusive, include increased GABA-ergic tone, selective alterations of the blood-brain barrier permeability and changes in neurotransmitter systems. The broad spectrum of symptoms in HE include forgetfulness, confusion, disorientation, concentration and memory problems, changes in mood, decreased alertness and responsiveness, changes in sleep habits, muscle tremors and stiffness, speech impairments, uncontrollable movements, agitation (Ferenci et al., 2002).

The diagnosis of HE is essentially based on clinical history and laboratory findings such as elevated ammonia levels. Additionally, specialized psychometric tests such as the number connection test (NCT), Digit Symbol Test (DST) and Psychometric Hepatic Encephalopathy Score (PHES) have been used in quantifying the minor deficits that may be present in patients with early HE.

Minimal hepatic encephalopathy (MHE) is a category of early HE without any overt neuropsychiatric symptoms but with subtle cognitive deficits (Ferenci et al., 1998). It is a common complication of cirrhosis and has been reported in 20% to 74% of patients (Dhiman et al., 2010), depending on the test used for diagnosis. It results in deficits in specific cognitive domains such as attention, vigilance, response inhibition, executive function and prospective memory. These deficits are often not apparent from a routine neurological exam or MMSE but can be detected on psychometric testing. The prompt identification and treatment of MHE are essential because MHE predicts progression to overt HE and impairs the capacity to drive which can have a significant impact on patients' quality of life (Romero-Gomez et al., 2001; Wein et al, 2004) .

Treatment of HE with or without liver transplantation has been shown to reverse the cognitive deficits and improve quality of life (Prasad et al., 2007; Sidhu et al., 2011). Although the PHES and NCT are the gold standard for diagnosing MHE, their utility is limited due to expensive copyright, a need for trained psychologists and the lack of reimbursements from insurance companies. A simpler test would therefore be beneficial to internists who could easily implement it in the clinic setting.

The inhibitory control task (ICT) is a computerized psychometric test that has been introduced recently as a diagnostic tool for MHE. It measures the ability to sustain attention and to inhibit responses to relevant stimuli, 2 basic cognitive domains that are impaired in MHE. During the ICT, the patient is presented with a continuous stream of letters at 500-ms intervals and interspersed within these letters are the letters X and Y. Subjects are instructed to only respond when the letters "X" and "Y" are alternated (called targets), independent of the letters between them. In contrast, patients are instructed to refrain from responding, i.e. inhibit their response, when "X" and "Y" are not alternating (called lures). Higher rates of target response, lower rates of lure response and shorter reaction times indicate better attention and response inhibition. One study by Bajaj et al. (2008) showed the ICT to be a reliable test with 87% sensitivity for the diagnosis of MHE, with MHE patients having higher ICT lures and lower targets compared to patients without MHE.

Patients with MHE have deficits in attention and prospective memory which are cognitive domains that are important to activities such as driving. Sustaining attention is important for learning and remembering new information, for e.g. keeping the car within the lane while driving and paying attention to pedestrians and cyclists. Prospective memory involves both working memory (to formulate, initiate, and modify plans of action) and retrospective memory (to recall what needs to be done at a particular time or in response to an external cue), for instance, remembering the correct exit while driving on the highway. The act of driving requires the ability to sustain attention and utilize prospective memory under stressful conditions. Impairment in any of these areas may result in serious consequences for patient with chronic liver disease, such as cirrhosis. Indeed, some studies of cirrhotic patients have shown that those with MHE have a diminished ability to drive and significantly more motor vehicle crashes and traffic violations than those without MHE (Bajaj et al., 2007, 2009). The reasons behind this are thought to be not only the obvious cognitive deficits, but also a greater tendency to fatigue at the wheel and poor insight into the cognitive deficiencies (Kircheis et al., 2009). In fact, driving simulator tests and questionnaire surveys have shown that patients with MHE who have been diagnosed using the ICT have impaired navigational skills and significantly higher crash rates (Bajaj et al., 2008, 2009).

In addition to the potential value of the ICT in detecting MHE, the test may be useful in uncovering temporary insults to attention and working memory that may arise in the presence of external stimuli such as music. Listening to music while driving is a pervasive practice and the relationship between background music and driving performance has been studied in the past (Unal et al., 2012; van der Zwaag et al., 2012). However these studies did not specifically address patients with cirrhosis, who are a population at higher risk of traffic accidents. The hypothesis of our study are (1) cirrhotic patients with MHE are expected to have lower ICT scores than patients without MHE and (2) these deficits are expected to worsen in the presence of music, suggesting music as a possible factor that could contribute to impaired attention and working memory, and hence impaired driving ability in cirrhotic patients. To this end, various types of music, including classical and heavy metal, will be used as a means of distracting cirrhotic patients while they are administered the ICT, to determine if there is any effect of listening to music on ICT scores. In addition to the ICT, the Digit Symbol Test, Number Connection Test, Cambridge Prospective Memory Test (CAMPROMPT), Stroop test, Fisk Fatigue Impact Scale and Epworth Sleepiness Scale will also be administered to quantify the degree of HE. While the use of ICT may not be appropriate for definitively predicting driving fitness, it may be valuable in uncovering deficits in attention and memory that arise while listening to music, which may ultimately aid in the counseling and education of patients regarding safe driving practices.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patient with cirrhosis
* Able to provide informed consent

Exclusion Criteria:

* History of alcohol abuse within six months
* Active gastrointestinal bleeding
* Unable to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least fifty subjects will be included in this study, including screening failures. There will be an equitable inclusion of both men and women in this study. Subjects must be between the ages of 18 and 70 to participate in this study. There is no restriction on race or ethnicity in this study. An effort will be made to recruit a diverse sample of participants.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Lure Response Inhibition on Inhibitory Control Test | The ICT will be administered with and without background music during a single visit.

SECONDARY OUTCOMES:
Target Responses on Inhibitory Control Test | The ICT will be administered with and without background music during a single visit.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Sigal, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Medical Center, New York, New York, United States